CLINICAL TRIAL: NCT00706225
Title: An Open-Label, Single/Multiple Dose, Non-Randomized, 3-Period, Crossover Study To Determine The Potential Drug Interaction Of Bazedoxifene On Conjugated Estrogens (CE) In Healthy Postmenopausal Women
Brief Title: Study Evaluating Potential Drug Interaction Of Bazedoxifene & Premarin In Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3115A1-1134
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Postmenopause
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Bazedoxifene and Conjugated Estrogens (BZA & CE)
  Interventions: Drug: Bazedoxifene and conjugated estrogens

INTERVENTIONS:
Drug: Bazedoxifene and conjugated estrogens — Bazedoxifene 20 mg tablet once daily for 7 days. Conjugated Estrogens 0.625 mg tablet, single doses one week apart.

SUMMARY:
Bazedoxifene (BZA) 20 mg tablet is an investigational medication (not approved by FDA) which is being studied for possible prevention and treatment of postmenopausal osteoporosis.

PREMARIN® (conjugated estrogens [CE]) is approved by FDA to treat moderate to severe symptoms of menopause (i.e., hot flashes, and/or vulvar and vaginal atrophy) and for the prevention of postmenopausal osteoporosis.

The purpose of this study is to evaluate the pharmacokinetics (absorption, distribution, breakdown and elimination in the body) of a single dose of PREMARIN® when administered together with multiple doses of bazedoxifene (BZA) to healthy postmenopausal women.

Information will also be obtained regarding the safety and tolerability of the study medications when given together to healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, postmenopausal woman, (either naturally or surgically and have blood hormone levels consistent with a postmenopausal state for specified subjects) between the ages of 35 and 70 years, inclusive
* Have not participated in a clinical drug study for at least 30 days prior to study medication administration,
* Must not have a history of drug or alcohol abuse within 1 year and do not consume more than 2 standard units per day of alcohol (a standard unit equals 12 ounces of beer, 1 ½ ounces of 80-proof alcohol or 6 ounces of wine)
* Must either be a non-smoker or smoke less than 10 cigarettes per day, and must be able to abstain from smoking during clinic confinements,
* Must not donate any other plasma or blood during the total study.
* All test results and study criteria for the study are met.

Exclusion Criteria:

* Only healthy postmenopausal women are eligible.
* Health assessed by clinical chemistry laboratory results and physical exam.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential pharmacokinetic (PK) interaction of multiple oral doses of bazedoxifene (BZA) and a single dose of conjugated estrogens (CE) when co administered to healthy postmenopausal women. | 3 months

SECONDARY OUTCOMES:
To assess the safety of conjugated estrogens (CE) and bazedoxifene (BZA) when co administered to healthy postmenopausal women. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Daytona Beach, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3115A1-1134&StudyName=Study%20Evaluating%20Potential%20Drug%20Interaction%20Of%20Bazedoxifene%20%26%20Premarin%20In%20Healthy%20Postmenopausal%20Women